CLINICAL TRIAL: NCT05326711
Title: Effects of Telerehabilitation-Based Motor Imagery Training on Pain in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Assoc Prof, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/29-24
Record Dates: First submitted 2021-11-16; First posted 2022-04-13 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis; Pain
Keywords: multiple sclerosis; motor imagery; pain; telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation-based motor imagery training (Experimental): The first 2 weeks of the treatment period, will reserved for implicit motor imagery / lateralization training. It will be performed by the "noi group application" application that can be downloaded to the participants' mobile devices. Participants will be asked to use the app 3 times a day. In each application session, the right / left discrimination of the region in the photograph will be requested within 5 seconds and 30 photographs will be shown for each painful region. Each session will last 2-3 minutes on average. For 3rd to 8th weeks of the treatment period telehabilitation-based motor imagery training will be given to the participants individually, in synchronization, using the Google Meet videoconference platform, under the guidance of a physiotherapist. The duration of the sessions will last 20-30 minutes.
  Interventions: Behavioral: Telerehabilitation-based motor imagery training
- Control (No Intervention): No specific intervention

INTERVENTIONS:
Behavioral: Telerehabilitation-based motor imagery training — Telerehabilitation has been defined as "the delivery of rehabilitation services through information and communication technologies".
  Arms: Telerehabilitation-based motor imagery training

SUMMARY:
In this studly, the effects of an 8-week telerehabilitation-based motor imagery training on pain and related factors in persons with multiple sclerosis will be investigated.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, progressive, and demyelinating disease of the central nervous system that affects more than 2.5 million people worldwide and is more common in young adults. The most common clinical signs and symptoms include motor dysfunction, fatigue, spasticity, cognitive impairment, depression, decreased quality of life, bladder and bowel dysfunction and pain. People with Multiple Sclerosis (pwMS) show a wide range of pain symptoms, from acute pain symptoms to chronic pain symptoms. Pain is an important symptom in pwMS and is often associated with disability. Pain is a fairly common symptom in pwMS. The prevalence of pain in MS was found to be 63%. In addition, 30% of pwMS describe pain as their most severe symptom.

In the studies, it was found that motor imagery training, which is defined as imagining movement without revealing the movement in reality, is a training at the cortical level and reduces pain by creating positive effects on the impaired body schema perception. However, the effect of motor imagery training on pain in pwMS has not been investigated before.

For this reason, the aim of this study is to investigate the effect of telerehabilitation-based motor imagery training protocol, guidance of a physiotherapist, on pain, fatigue, anxiety, depression, quality of life and sleep quality in pwMS.

Persons who followed by the outpatient Multiple Sclerosis Clinic of Dokuz Eylül University Hospital will participate in the study. A total of 32 participants will randomly be divided into 2 groups. (1) Telerehabilitation-based motor imagery training, (2) Control group. Telerehabilitation-based motor imagery training group will individually receive telerehabilitation-based motor imagery training under the guidance of a physiotherapist for 8 weeks.

The first 2 weeks of the treatment period, will reserved for implicit motor imagery / lateralization training. It will be performed by the "noi group application" application that can be downloaded to the participants' mobile devices (smartphone or tablet). Lateralization training will be aimed at the initially evaluated areas of the participants (neck, back, shoulder, knee, hand/wrist, foot/ankle) that have a pain level of at least 30 mm according to the Visual Pain Scale (VAS). In the application, the participants will be asked to discriminant right and left with simple photographs of the painful areas determined at the beginning, and more complex photographs will be used as the training progresses. Participants will be asked to use the app 3 times a day. In each application session, the right / left discrimination of the region in the photograph will be requested within 5 seconds and 30 photographs will be shown for each painful region. Each session will last 2-3 minutes on average, depending on the number of painful areas of the participants. Controls will be made over the results sent to the e-mail address of the physiotherapist through the application. For 3rd to 8th weeks of the treatment period telehabilitation-based motor imagery training will be given to the participants individually, in synchronization, using the Google Meet videoconference platform, under the guidance of a physiotherapist. Participants will participate the treatment with their smart phones, tablets or computers that have an active internet connection and are suitable for meeting via videoconference. The duration of the sessions will last 20-30 minutes.

The control group will not receive treatment other than their routine treatment, and the patients will be informed that the control group participants will be treated if the participants wish at the end of the study. The assessments will be applied at baseline, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with MS according to McDonald diagnostic criteria
* Not having an attack in the last 3 months.
* To have sufficient smartphone/tablet or computer knowledge to participate in the study or to have a relative who can help in this regard.
* Having an active internet connection at home.
* Having a smart phone/tablet or computer suitable for videoconferencing.
* Having a smartphone or tablet.
* Having a pain level of at least 30 mm on the 100 mm visual analog scale (VAS) for at least 3 months in at least one of the hand/wrist, foot/ankle, knee, shoulder, neck and back regions.
* No change in medications used for pain in the last 2 months.
* Not receiving additional treatment other than routine treatments.
* To be able to read and understand Turkish.

Exclusion Criteria:

* Pregnancy
* Having a musculoskeletal, cardiovascular, pulmonary, metabolic, or other disease severe enough to preclude participation in the study.
* Presence of conditions other than MS that can cause pain, such as cancer, diabetes, overt osteoarthritis, or rheumatoid arthritis based on laboratory or imaging findings
* Having a psychiatric illness.
* Presence of severe cognitive impairment detected by the physician at a level that prevents the tests from being performed
* Having severe vision and hearing problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Score | The assessments will be applied at baseline, 8, and 12 weeks.
  VAS will be used to numerically determine the general pain intensities felt by participants in the last 2 days and the pain intensities of the areas they feel painful on six regions: neck, shoulder, back, hand/wrist, knee, foot/ankle. Participants will be told that 0mm above the 100mm line had "no pain"; It will be stated that 100 mm represents "the most unbearable pain". The degree of pain will be recorded numerically between 0 and 100.

SECONDARY OUTCOMES:
Expanded Disability Status Scale | The assessment will be applied at baseline.
  Expanded Disability Status Scale is the most frequently used scale in evaluating the disability of pwMS. Scoring based on neurological examination findings takes a value between 0-10. While 0 shows normal neurological findings, 10 means death due to MS. In this scale in which pyramidal, cerebral, cerebellar, visual, sensory, brainstem, bladder and bowel functions are scored, the best performance of the patient without any special effort is evaluated.
Change in Patient-Determined Disease Steps Scale Score | The assessments will be applied at baseline and 8 weeks.
  Patient-Determined Disease Steps Scale was designed in 1995 as a self-reported outcome measure to enable neurologists without EDSS evaluator certification to measure the level of disability of pwMS. It consists of one question. In PDDS, the patient is asked to choose one of the 9 items that best describes his current walking ability.
Change in Numeric Rating Scale Score | The assessments will be applied at baseline, 8, and 12 weeks
  Numeric Rating Scale will be used to determine pain levels in functional activities of participants. Participants are asked to name the number representing the amount of pain, where 0 is "no pain" and 10 is "most unbearable pain". Participants will be asked to identify the 5 activities they find most difficult to do because of their pain and to evaluate their pain for activities.
Change in PainDETECT Questionnaire Score | The assessments will be applied at baseline, 8, and 12 weeks
  PainDETECT Questionnaire is used to determine neuropathic pain of participants. The questionnaire assesses the typical symptoms, signs, and extent of pain of neuropathic pain. A questionnaire score of ≥19 indicates probable neuropathic pain, a score of 13 to 18 indicates that the result is uncertain, and neuropathic pain of ≤12 is unlikely.
Change in Nordic Musculoskeletal Questionnaire Score | The assessments will be applied at baseline, 8, and 12 weeks
  Nordic Musculoskeletal Questionnaire is used to determine the musculoskeletal system pain of participants. Questionnaire; whether there is pain on a figure showing the nine regions anatomically: neck, shoulder, back, elbow, hand/wrist, waist, hip/thigh, knee, foot/ankle, whether you have experienced pain in the last week or one year. questions whether the pain affects work/home life. The form consists of three parts and provides descriptive information about whether the participants have experienced various musculoskeletal pain in the last year and in the last seven days, and whether these pains affect their work/home life. The classical evaluation method is in the form of calculating the response distribution ratios and obtaining descriptive data.
Change in Kinesthetic and Visual Imagery Questionnaire- 20 Score | The assessments will be applied at baseline, 8, and 12 weeks.
  Kinesthetic and Visual Imagery Questionnaire- 20 is used to determine the motor imagery skills of participants. The questionnaire consists of a total of 10 movements measuring 5 visual and 5 kinesthetic visualization skills developed to determine the extent to which individuals visualize and feel the imagined movements. The participant give a score between 1 and 5, as "1 point: no image, 5 points: as clear as the original" for the image in the imagery. At the end of the questionnaire, visual imagery score, kinesthetic imagery score and total score are calculated.
Change in Modified Fatigue Impact Scale Score | The assessments will be applied at baseline, 8, and 12 weeks
  Modified Fatigue Impact Scale is used to determine the fatigue level of participants. The questionnaire consists of a total of 21 questions evaluating the physical, cognitive and psychosocial effects of fatigue. Each item is given a score of 0-4. Low score indicates a low degree of fatigue
Change in Multiple Sclerosis İnternational Quality of Life Questionnaire Score | The assessments will be applied at baseline, 8, and 12 weeks.
  Multiple Sclerosis İnternational Quality of Life Questionnaire is used to determine the quality of life of participants. The questionnaire is a self-filled 31-item scale measuring health-related quality of life. The questionnaire questions quality of life in various areas, including activities of daily living, psychological well-being, symptoms, relationships with friends, relationships with family, health care team satisfaction, emotional life and sex life, coping and rejection. The total score is between 0 and 100, and high scores indicate high quality of life perception
Change in Pittsburgh Sleep Quality Index Score | The assessments will be applied at baseline, 8, and 12 weeks.
  Pittsburgh Sleep Quality Index is used to determine the sleep quality of participants. The questionnaire includes 24 questions evaluating the sleep quality of the participants for the last month. 19 of these are self-report questions and are answered by the participants themself. Five questions are answered by the participant's spouse or roommate and are used for clinical information only, not included in scoring. The total score takes a value between 0 and 21. Sleep quality of those with a total score of 5 or less was "good"; Those with a score above 5 are considered to have "poor" sleep quality.
Change in Epworth Sleepiness Scale Score | The assessments will be applied at baseline, 8, and 12 weeks.
  Epworth Sleepiness Scale is used to determine the daytime sleepiness of participants. The scale consists of 8 items. The score of each item varies between 0-3 and the total score varies between 0-24. High scores indicate high daytime sleepiness
Change in Hospital Anxiety and Depression Scale (HADS) Score | The assessments will be applied at baseline, 8, and 12 weeks
  HADS is used to determine the risk of anxiety and depression in the participants and to measure its level and severity. It is a self-report scale consisting of 7 anxiety and 7 depression related questions in total and two subscales. Items are scored with a 3-level Likert-type scale. High scores indicates high anxiety and depression level.
Change in Mental Chronometer Time Ratio for Timed Up and Go Test Score | The assessments will be applied at baseline, 8, and 12 weeks
  Mental Chronometer Time measurement will be performed with the Timed Up and Go Test. During the Timed Up and Go Test, the participants will be asked to get up from a chair, walk three meters, turn around the board at the end of 3 meters, walk back to the chair and sit. After imagining the movement during the test, participants will actually apply the test. The temporal coherence between real and imagined motion will be calculated in terms of delta time with the formula "(real motion-imagined motion)/[(actual motion + imagined motion)/2] x 100". The duration of actual and imagined movements will be recorded with an electronic stopwatch. The time during the actual movement will be recorded by the physiotherapist. The imaginary time will be recorded by the participants. The participants will start the stopwatch when they started to move the imagined movement and will stop it when the participants completed the imagined movement. Closer scores to 100 mean better temporal coherence.
Change in California Verbal Learning Test-II Score | The assessments will be applied at baseline, 8, and 12 weeks
  The California Verbal Learning Test-II is used to assess verbal memory. Higher scores indicate better verbal memory.
Change in Revised Brief Visuospatial Memory Test Score | The assessments will be applied at baseline, 8, and 12 weeks
  The Revised Brief Visuospatial Memory Test is used to assess visuospatial memory. Higher scores indicate better visuospatial memory.
Change in Symbol Digit Modalities Test Test Score | The assessments will be applied at baseline, 8, and 12 weeks
  The Symbol Digit Modalities Test is used to assess information processing speed. Using a reference key, the test taker has 90 seconds to pair specific numbers with given geometric figures in the Symbol Digit Modalities Test. The correct matches are calculated as the test score. Higher scores indicate better information processing speed.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir, Inciralti
  - Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir